CLINICAL TRIAL: NCT04493099
Title: A Phase 1/2 Study of Alvocidib in Combination With Decitabine and Venetoclax in Patients With Relapsed or Refractory AML or as Frontline Therapy in Unfit Patients With AML
Brief Title: Alvocidib in Combination With Decitabine and Venetoclax in Patients With Relapsed or Refractory AML or as Frontline Therapy in Unfit Patients With AML
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The original sponsor was acquired by a new company and has elected to end funding for all Investigator Sponsored Trials (ISTs)
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-1053; NCI-2020-05266 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-1053 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-27; First posted 2020-07-30 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — cytokine inducible SH2-containing protein; alvocidib; Decitabine; Injections; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, alvocidib hydrochloride, venetoclax) (Experimental): INDUCTION: Patients receive decitabine IV over 1 hour on days 1-10, alvocidib hydrochloride IV over 1 hour on days 1-3, 1-5, 1-7, 1-10, or 1-14, and venetoclax PO QD on days 1-14 in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION: Patients receive decitabine IV over 1 hour on days 1-5, alvocidib hydrochloride IV over 1 hour on days 1-3, 1-5, 1-7, 1-10 or 1-14, and venetoclax PO QD on days 1-10. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Alvocidib Hydrochloride; Drug: Decitabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Alvocidib Hydrochloride — Given IV
  Other Names: 4H-1-Benzopyran-4-one, 2-(2-chlorophenyl)-5, 7-dihydroxy-8-(3-hydroxy-1-methyl-4-piperidinyl)-, hydrochloride, (-)-cis-; Flavopiridol Hydrochloride; HL-275; HMR 1275; L-86-8275; L-868275; MDL 107,826A; MDL-107826A
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2''-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Drug: Venetoclax — Given PO
  Other Names: ABT-0199; ABT-199; ABT199; GDC-0199; RG7601; Venclexta; Venclyxto

SUMMARY:
This phase I/II trial investigates the side effects and best dose of alvocidib when given together with decitabine and venetoclax and to see how well it works in treating patients with acute myeloid leukemia that has come back (relapsed), has not responded to previous treatment (refractory), or as frontline treatment for patients unable to receive other therapies (unfit). Alvocidib, decitabine, and venetoclax may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of alvocidib hydrochloride (alvocidib) in combination with decitabine and venetoclax in relapsed or refractory patients with acute myeloid leukemia (AML) or as frontline therapy in unfit/frail patients with AML. (Phase I) II. To determine the efficacy alvocidib in combination with decitabine and venetoclax in relapsed or refractory patients with acute myeloid leukemia (AML) or as frontline therapy in unfit/frail patients with AML. (Phase II)

SECONDARY OBJECTIVE:

I. To determine the preliminary assessment of efficacy by response to revised International Working Group (IWG) criteria and time to response variables, including overall survival (OS), event-free survival (EFS) and duration of response (DOR) of patients treated with this combination.

EXPLORATORY OBJECTIVES:

I. To determine the minimal residual disease (MRD) after treatment with this combination and its impact in long-term outcome.

II. To determine the effect of the level of pre-treatment expression of BCL-2 and MCL-1 (by BH3 profiling) with response to this combination.

III. To determine the effect of this treatment combination on responding patients transitioning to hematopoietic stem cell transplantation (HSCT).

OUTLINE: This is a phase I, dose-escalation study of alvocidib followed by a phase II study.

INDUCTION: Patients receive decitabine intravenously (IV) over 1 hour on days 1-10, alvocidib hydrochloride IV over 1 hour on days 1-3, 1-5, 1-7, 1-10, or 1-14, and venetoclax orally (PO) once daily (QD) on days 1-14 in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION: Patients receive decitabine IV over 1 hour on days 1-5, alvocidib hydrochloride IV over 1 hour on days 1-3, 1-5, 1-7, 1-10 or 1-14, and venetoclax PO QD on days 1-10. Treatment repeats every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsed or refractory acute myeloid leukemia by World Health Organization (WHO) criteria. Unfit/frail patients with newly diagnosed AML are also eligible if not considered good candidates to receive a higher intensity therapy

  * A patient is considered unfit or frail if has three or more of the five factor below:

    * Unintentional weight loss of 10 pounds or more in a year
    * General feeling of exhaustion
    * Weakness as measured by grip strength
    * Slow walking speed
    * Low levels of physical activity
* Eastern Cooperative Oncology Group (ECOG) performance status score of =< 3
* Total serum bilirubin =< 2 x upper limit of normal (ULN). Patients with known Gilbert's syndrome may have a total bilirubin up to =< 3 x ULN
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) =< 3 x ULN; or =< 5 x ULN in case of suspected leukemic liver involvement
* Serum creatinine =< 2.0 mg/dl
* Females of childbearing potential must have a negative serum or urine beta human chorionic gonadotropin (B-HCG) pregnancy test result within 1 week (+/-3 days) prior to the first dose of study drugs and must agree to use one of the following effective contraception methods during the study and for 30 days following the last dose of study drug. Effective methods of birth control include:

  * Birth control pills, shots, implants (placed under the skin by a health care provider) or patches (placed on the skin)
  * Intrauterine devices (IUDs)
  * Condom or occlusive cap (diaphragm or cervical/vault caps) used with spermicide
  * Abstinence
  * Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation, oophorectomy, and/or hysterectomy
* Males who have partners of childbearing potential must agree to use an effective contraceptive method (such as condom used with spermicide or abstinence) during the study and for 30 days following the last dose of study drug
* Patients or their legally authorized representative must provide written informed consent

Exclusion Criteria:

* Patients with t(15;17) karyotype abnormality or acute promyelocytic leukemia
* History of another primary invasive malignancy that has not been definitively treated and in remission. Patients with non-melanoma skin cancers or with carcinomas in situ are eligible regardless of the time from diagnosis (including concomitant diagnoses)
* Presence of clinically significant uncontrolled central nervous system (CNS) pathology such as epilepsy, childhood or adult seizure, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
* Evidence of active cerebral/meningeal disease. Patients may have history of CNS leukemic involvement if definitively treated with prior therapy and no evidence of active disease at the time of consent with at least 2 consecutive spinal fluid negative assessments for residual leukemia and negative imaging (imaging required only if previously showing evidence of CNS leukemia not otherwise documented by spinal fluid assessment)
* Patients with active unstable angina, concomitant clinically significant active arrhythmias, myocardial infarction within 6 months, or congestive heart failure New York Heart Association class III-IV. Patients with a cardiac ejection fraction (as measured by either multigated acquisition scan [MUGA] or echocardiogram) < 45% are excluded
* Patients with uncontrolled, active infections (viral, bacterial, or fungal)
* Known active hepatitis B or C infection, or known seropositivity for human immunodeficiency virus (HIV)
* Patients with liver cirrhosis or other serious active liver disease or with suspected active alcohol abuse
* Allogeneic hematopoietic cell transplantation (HSCT) within 6 months before the start of protocol-specified therapy, or with active acute/chronic graft-versus-host disease (GvHD) requiring systemic treatment; or receiving immunosuppression for GvHD prophylaxis within 2 weeks from the start of study therapy
* Prior chemotherapy/radiotherapy/investigational therapy within 2 weeks before the start of study drugs with the following exception:

  * To reduce tumor burden, leukocytosis (circulating blast count) or palliation: Intravenous cytarabine and/or hydroxyurea. No washout is necessary for these agents. Patients must have recovered from acute non hematologic toxicity (to =< grade 1) of all previous therapy prior to enrollment
* Females who are pregnant or lactating
* Male or female subjects of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with institution's standards
* Other severe, uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and/or would make the patient inappropriate for enrollment into this study
* Prior treatment with alvocidib

  * Prior use of venetoclax single agent or any venetoclax-based combination therapy is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-10-12 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
Overall incidence and severity of all adverse events (Phase I) | Up to 6 years
  Measured using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Overall response rate (ORR) (Phase II) | Up to 6 years
  Will estimate the response rate for the combination treatment, along with the 95% credible interval.

SECONDARY OUTCOMES:
Duration of response | Up to 6 years
  The duration of response is defined as the number of days from the date of initial response (partial response [PR] or better) to the date of first documented disease progression/relapse or death, whichever occurs first.
Event free survival | Up to 6 years
  Event-free survival is defined as the number of days from the date of treatment initiation (e.g., cycle 1 day 1 [C1D1]) to the date of documented treatment failure, relapses from complete response (CR), or death from any cause, whichever occurs first, and will be calculated for all patients. Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.
Overall survival | From treatment start till death or last follow-up, assessed up to 6 years
  Will be estimated using the method of Kaplan and Meier. Comparisons of time-to-event endpoints by important subgroups will be made using the log-rank tests.

CONTACTS AND LOCATIONS:
Overall Officials: Yesid Alvarado-Valero, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: http://www.mdanderson.org — http://www.mdanderson.org